CLINICAL TRIAL: NCT05119998
Title: A Phase I, Open-label, Multicenter, Dose-escalation Study Evaluating the Safety, Tolerability, and Potential Efficacy of IBI325, an Anti-CD73 Antibody, in Patients With Advanced Solid Tumor
Brief Title: A Phase I Study of IBI325 in Patients With Advanced Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI325A101
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2022-10

CONDITIONS: Solid Tumor
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI325 and sintilimab combination does-escalation (Experimental)
  Interventions: Drug: IBI325 + sintilimab
- IBI325 monotherapy does-escalation (Experimental)
  Interventions: Drug: IBI325

INTERVENTIONS:
Drug: IBI325 + sintilimab — IBI325 + sintilimab combination does-escalation Patients will receive IBI325 and sintilimab until progressive disease, intolerability, or other reasons leading to treatment discontinuation
  Arms: IBI325 and sintilimab combination does-escalation
Drug: IBI325 — IBI325 monotherapy does-escalation Patients will receive IBI325 until progressive disease, intolerability, or other reasons leading to treatment discontinuation
  Arms: IBI325 monotherapy does-escalation

SUMMARY:
The primary objective of this phase I study is to evaluate the safety and potential efficacy and to determine the recommended phase 2 dose (RP2D) of IBI325 in patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, locally advanced unresectable or metastatic tumors.
2. At least one evaluable or measurable lesion per RECIST 1.1
3. Male or female subject at least 18 years old and no more than 75 years old.
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) performance status 0 or 1.
5. Must have adequate organ function
6. Be able to provide archived or fresh tumor tissues-

Exclusion Criteria:

1. Previous exposure to any anti-CD73 monoclonal antibody
2. Subjects participating in another interventional clinical study, except for during the survival follow-up phase of the studies.
3. Unstable central nervous system netastases
4. Known active autoimmune disease or inflammatory disease
5. Known active infectious disease
6. Other uncontrolled systematic disease that may increase the risk of participating the study-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with DLT | 28 days post first dose
  Number of patients who experienced a dose-limiting toxicity within the first 28 days after the first dose
Number of patients with treatment related AEs | Up to 90 days post last dose
  Number of patients who experienced a treatment related AEs from the first dose until 90days after the last dose

SECONDARY OUTCOMES:
Number of patients with response | Every 6 weeks until progressive disease or up to 24 months after treatment
  Number of patients with response per RECIST 1.1
The area under the curve (AUC) | Up to 90 days post last dose
Maximum concentration (Cmax) | Up to 90 days post last dose
Time at which maximum concentration (Tmax) | Up to 90 days post last dose
The half-life (t1/2) | Up to 90 days post last dose
Positive rate of ADA and Nab | Up to 90 days post last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Province Cancer Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No